CLINICAL TRIAL: NCT05116345
Title: DEXTENZA for the Treatment of Pain and Inflammation Following Surgical Trabeculectomy and Ahmed Valve Procedures
Acronym: DEXTenSiVe
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brian Jerkins, MD (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Brian Jerkins, MD, Assistant Professor, University of Tennessee
Organization: University of Tennessee (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The DEXTenSiVe Study
Record Dates: First submitted 2021-10-26; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Glaucoma Following Surgery
MeSH Terms: interventions — Calcium Dobesilate; Dexamethasone; Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEXTENZA (Experimental): a single intracanalicular dexamethasone (0.4 mg) insert
  Interventions: Drug: DEXTENZA
- Topical Dexamethasone Treatment (Active Comparator): Standard of care topical dexamethasone treatment through Month 2 dosing and tapering following:
  6x/day week 1 4x/day weeks 2-4 2x/day weeks 5-8 Day of surgery dexamethasone ointment and patch will be applied post-surgically for overnight treatment and removed at post-operative day 1 visit in Group B eyes.
  Interventions: Drug: Topical Dexamethasone

INTERVENTIONS:
Drug: DEXTENZA — Intracanalicular Dexamethasone ophthalmic insert (0.4mg)
  Other Names: Dexamethasone (0.4mg) Insert
  Arms: DEXTENZA
Drug: Topical Dexamethasone — topical dexamethasone drops
  Arms: Topical Dexamethasone Treatment

SUMMARY:
This is a prospective, comparative, open-label, single-center, randomized, investigator-sponsored clinical study and seeks to investigate clinical outcomes with standard of care and high dose DEXTENZA treatment compared to standard of care topical dexamethasone in patients undergoing trabeculectomy, trabeculectomy Ex-PRESS, Xen Gel stent, and Ahmed Valve surgery. Patients will be followed through 6 months. After screening a given patient for inclusion and exclusion criteria, and gaining informed consent, eyes of n=30 patients will be randomized to one of the following two groups (n=15per group) and followed from Baseline through Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed written consent prior to participation in any study-related procedures
* Patient is diagnosed with glaucoma and undergoing trabeculectomy, trabeculectomy Ex-PRESS, Xen Gel stent, or Ahmed Valve surgery

Exclusion Criteria:

* Have used topical corticosteroid treatment up to 48 hours prior to the baseline visit
* Have used oral corticosteroid within the past 14 days prior to baseline visit (Patients using stable doses of inhaled corticosteroids for 30 days prior to baseline visit can be included in the study)
* Have received intravitreal or sub-Tenon corticosteroid treatment prior to baseline visit or Ozurdex ® in the study eye within the 6 months prior to the baseline visit
* Are currently using prescribed nonsteroidal anti-inflammatory agents or prescribed immunosuppressive agents, unless the dose has been stable for the last 6 weeks and no change in dosing is anticipated for the duration of the study
* Are pregnant or lactating female, or female of childbearing age using inadequate birth control method
* Have participated in another investigational device or drug study within 30 days of the baseline visit
* Anterior chamber cells present at time of enrollment
* Known allergy to dexamethasone or prednisolone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Mean change in intraocular pressure (IOP) | From baseline through month 6
  mean change in intraocular pressure (IOP) from day of surgery and proportion of eyes requiring additional topical dexamethasone or anti-metabolite therapy over time

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) | From baseline through month 6
  Mean change in BCVA using Snellen eye charts
Mean change in Visual Field (MD) | From baseline through month 6
  Mean change in Visual Field (MD) will be detected using a perimeter device. The patient looks into the perimeter at a center target. Only one eye is tested at a time. The eye not being tested is covered with an eye patch. Small, dim lights will flash in the device and the patient will press a button each time they see the light. The results will show if the patient has had any changes in their visual field.
Conjunctival healing outcomes as defined by proportion of eyes requiring needling intervention associated with scar/fibrin development | From baseline through month 6
  Conjunctival healing outcomes as defined by proportion of eyes requiring needling intervention associated with scar/fibrin development
Proportion of eyes with absence of anterior chamber (AC) cells (score of 0) as measured by the Standardization of Uveitis Nomenclature (SUN) scale | From baseline through month 6
  Proportion of eyes with absence of anterior chamber (AC) cells (score of 0) as measured by the Standardization of Uveitis Nomenclature (SUN) scale
Time to resolution of anterior chamber (AC) cells and/or AC flare | From baseline through month 6
  Time to resolution of anterior chamber (AC) cells and/or AC flare
Proportion of eyes with absence of pain as measured by pain scale of 1-10 (pain score of 0 = absence) | From baseline through month 6
  Proportion of eyes with absence of pain as measured by pain scale of 1-10 (pain score of 0 = absence)
Number of patient call backs to medical staff regarding post-operative management of pain or medication management/dosing inquiry as documented by Electronic Health Record (E.H.R.). | From baseline through month 6
  Number of patient call backs to medical staff regarding post-operative management of pain or medication management/dosing inquiry as documented by Electronic Health Record (E.H.R.).
Incidence and severity of adverse events | From baseline through month 6
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jerkins, MD, Principal Investigator — University of Tennessee
Locations (1):
- Hamilton Eye Institute, Memphis, Tennessee, United States

REFERENCES:
- [Background] Okeke CO, Quigley HA, Jampel HD, Ying GS, Plyler RJ, Jiang Y, Friedman DS. Adherence with topical glaucoma medication monitored electronically the Travatan Dosing Aid study. Ophthalmology. 2009 Feb;116(2):191-9. doi: 10.1016/j.ophtha.2008.09.004. Epub 2008 Dec 12. PMID 19084273
- [Background] Lee A, Blair HA. Correction to: Dexamethasone Intracanalicular Insert: A Review in Treating Post-Surgical Ocular Pain and Inflammation. Drugs. 2020 Aug;80(12):1265. doi: 10.1007/s40265-020-01366-0. PMID 32700064